CLINICAL TRIAL: NCT02097160
Title: How Much Vitamin D is Needed in Milk Products to Support Vitamin D Intake and Bone Health in Children?
Acronym: D-KIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Hope Weiler, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: HW-14-01
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: childhood; healthy; vitamin D; bone; dairy products

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group 1 (Active Comparator): regular fortified milk + regular cheese/yogurt
  Interventions: Other: Control Group 1
- Intervention Group 2 (Experimental): Vitamin D fortified yogurt and cheese; vitamin D dose increment of 252 IU vs grp 1
  Interventions: Other: Vitamin D fortified yogurt and cheese products
- Intervention Group 3 (Experimental): Vitamin D fortified yogurt and cheese, vitamin D dose increment of 420 IU vs grp 1
  Interventions: Other: Vitamin D fortified yogurt and cheese products

INTERVENTIONS:
Other: Vitamin D fortified yogurt and cheese products
  Arms: Intervention Group 2; Intervention Group 3
Other: Control Group 1
  Arms: Control Group 1

SUMMARY:
The study is a parallel interventional randomized dose-response trial designed to improve vitamin D intakes through food in a group of healthy 2 - 7.9 year old children. Subjects will be recruited from the general population in the greater Montreal area. The study will be conducted at the Mary Emily Clinical Nutrition Research Unit of McGill University. Children will be required to attend two study visits. Some information will be collected through monthly telephone survey to the parents. The investigators will add vitamin D to cheese and yogurt for daily consumption at home over a three month period. All products will be provided to the parents in the form of coded containers that do not contain any labels aside from the group and expiration date. Ingredient lists will be provided upon consenting to the study. To better understand vitamin D status; dietary intake, hematology, serum biochemistry including 25(OH)D, growth, and body composition will be measured at the beginning and end of the three month study period. In addition, bone mass at baseline will be assessed. Sun exposure will be documented and a skin pigmentation test will be used to more objectively assess chronic sun exposure. The investigators will also investigate the association between vitamin D intake and status with immune function.

ELIGIBILITY:
Inclusion Criteria:

* Children will be pre-pubertal
* Healthy
* Regularly consume milk and milk products
* Healthy weights

All races will be studied.

Exclusion Criteria:

* Chronic diseases (including asthma) or medications known to affect vitamin D, infections or the immune system; known anaemia, small size at birth or preterm birth <37 wk gestation
* No milk allergy or lactose intolerance, no nutritional supplements Less than 1/3rd of preschool age children take a supplement based on our work; it will thus not be a limitation for recruitment to exclude supplement users. We will not study obese children since the response to exogenous vitamin D intervention is reduced.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
25(OH)D serum concentrations | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hope A Weiler, PhD, Principal Investigator — McGill University

REFERENCES:
- [Derived] Brett NR, Lavery P, Agellon S, Vanstone CA, Maguire JL, Rauch F, Weiler HA. Dietary vitamin D dose-response in healthy children 2 to 8 y of age: a 12-wk randomized controlled trial using fortified foods. Am J Clin Nutr. 2016 Jan;103(1):144-52. doi: 10.3945/ajcn.115.115956. Epub 2015 Dec 16. PMID 26675772